CLINICAL TRIAL: NCT06723327
Title: The Effect of Preoperative Culture Timing on Postoperative Outcomes of Retrograde Intrarenal Surgery
Status: Recruiting | Type: Observational
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Mehmet Fatih Şahin, Assistant Professor, Namik Kemal University
Other Study IDs: 2024.304.11.11
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Urinary Infections; Urolithiasis
Keywords: urine culture; urolithiasis; kidney stone; retrograde intrarenal surgery
MeSH Terms: conditions — Urolithiasis; Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine culture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with 2 sterile urine cultures: Before retrograde intrarenal surgery, patients with sterile urine culture 2 weeks before the surgery and morning urine culture
- Patients with only one sterile urine culture: Before retrograde intrarenal surgery, patients having sterile urine culture 2 weeks before the surgery and positive morning urine culture

SUMMARY:
The rate of complications (unexpected situations) after retrograde intrarenal surgery is reported to be 9-25%, and the majority of these are postoperative infections. Surgery must be performed under sterile (microbial-free) urine culture to prevent these complications. There are guideline recommendations regarding sterile urine culture reporting, but it is not clear how long in advance it should be taken. The possibility of the patient becoming infectious again during the period leading up to surgery is a condition that needs to be determined. Therefore, the culture taken before surgery should be compared with the urine culture result taken at the latest possible time before the operation.

DETAILED DESCRIPTION:
Retrograde Intrarenal Surgery (RIRC) (a surgery to fragment stones inside the kidney by entering from the distal end of the urinary tract with a camera system and light optical imaging device) is increasingly used today thanks to the developments in laser and scope (imaging device) technology. The risk of complications (unexpected situations) after this surgery is reported as 9-25%, most of which are infections. These infections can be severe conditions that can lead to septic shock (system failure due to severe infection) and death, as well as fever requiring only antipyretics (fever reducers).

Preventing infectious complications is as important as ensuring stone-free status for this surgery. For this purpose, surgery must be performed under sterile (microbe-free) urine culture. Patients with positive urine cultures should be taken to surgery due to increased pressure on the kidney, which can cause reflux (backflow of the kidney into the bloodstream) and infectious urine entering the circulation, leading to septicemia (microbes mixing into the bloodstream).

There are guideline recommendations regarding sterile urine culture reporting, but it is not clear how long in advance it should be taken. In the American Urology guidelines, a sterile urine culture within 1 month is sufficient to be taken to surgery, but no period is specified in the European Urology guidelines. The possibility of the patient becoming infected again during the period leading up to surgery is a condition that needs to be determined. Therefore, the culture taken before surgery should be compared with the urine culture result taken at the latest possible period before the operation. This study aims to evaluate the preoperative and morning urine culture results and compare the postoperative results of patients with this difference.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients who had a urine culture taken 2 weeks before the operation and reported as sterile

Exclusion Criteria:

* Patients under 18 years of age
* Patients without sufficient data
* Patients with a urine culture more than 2 weeks before retrograde intrarenal -surgery
* Patients with a positive urine culture before retrograde intrarenal surgery
* Patients with renal anatomic anomalies
* Patients with a solitary (single) kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort of 950 patients with two negative preoperative urine cultures and patients with 50 positive urine cultures on the operation morning.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative infection rates | within 2 weeks after the surgery
  Is there a difference in postoperative infectious complications between patients with two sterile preoperative urine cultures and patients with sterile cultures 2 weeks before the operation but positive urine cultures taken on the morning of the operation?

CONTACTS AND LOCATIONS:
Locations (1):
- Tekirdag Namık Kemal University, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mekayten M, Heifetz EM, Sompolinsky Y, Lorber A, Duvdevani M, Strahilevitz J. Timing of midstream urine culture before endourological procedure-can we do better?-A comparative study. Urolithiasis. 2023 Aug 27;51(1):110. doi: 10.1007/s00240-023-01483-x. PMID 37634153
- [Background] Akkas F, Cinislioglu N, Haciislamoglu A, Atar FA, Guner E, Karadag S. Does time elapsed between urine culture and retrograde intrarenal surgery affect the rate of systemic inflammatory response syndrome? Actas Urol Esp (Engl Ed). 2022 May;46(4):223-229. doi: 10.1016/j.acuroe.2022.02.003. Epub 2022 Feb 21. English, Spanish. PMID 35210199